CLINICAL TRIAL: NCT06199193
Title: Design of Personalised SupplemenTs Based on the Gut MicRobiota of Alzheimer Patients Through Network and Artificial Intelligence Analysis
Brief Title: Design of Personalised SupplemenTs Based on the Gut MicRobiota Through Artificial Intelligence for Alzheimer's Patients
Acronym: TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other); Universidad Europea de Madrid (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2021-123700OB-I00
Record Dates: First submitted 2023-12-05; First posted 2024-01-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Gut Microbiota
Keywords: Alzheimer's disease; Gut Microbiota; Physical exercise; Artificial intelligence; Supplementation
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Group 1: Control healthy humans with normal diet (n=30) Group 2: Alzheimer patients with normal diet (n=30). Group 3: Alzheimer patients with designed supplements(n=30)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Human patient (non-Alzheimer) with routine normal diet (No Intervention): Control human patients (60),non suffering from Alzheimer, will continue with their normal dietary habits and samples will be collected.
- Alzheimer patients with routine normal diet and dietary counseling (Sham Comparator): Alzheimer patients (60) will continue with their routine normal diet and samples will be collected.
  Interventions: Dietary Supplement: Dietary counseling
- Alzheimer patients with personalized diet (Experimental): Alzheimer patients (30) will be given personalized diet, with supplements based on the gut microbiota (elaborated through AI analyses) or a standard supplement (n=30) Samples will be collected.
  Interventions: Dietary Supplement: Personalized diet

INTERVENTIONS:
Dietary Supplement: Personalized diet — Personalized supplement designed by artificial intelligence based on the intestinal microbiota and incorporated into diets
  Arms: Alzheimer patients with personalized diet
Dietary Supplement: Dietary counseling — Dietary advice will be provided to adapt the diet to the nutritional objectives and recommended intakes.
  Arms: Alzheimer patients with routine normal diet and dietary counseling

SUMMARY:
Studies indicate that the intestinal microbiota could have an implication in Alzheimer's disease; recently, a positive relationship has been established between levels of bacterial lipopolysaccharide (LPS) and cerebral amyloidosis and a negative relationship between the production of the chain fatty acid cuts butyrate by the intestinal microbiota and cerebral amyloidosis. Currently there is no effective treatment for Alzheimer's, but studies indicate that a healthy diet such as the Mediterranean diet and physical exercise delay the symptoms of this disease. For all these reasons, it is postulated that introducing changes in the intestinal microbiota through diet may be a new treatment or serve as an adjuvant treatment for Alzheimer's disease.

DETAILED DESCRIPTION:
The study consists of three main stages, a first part in which healthy subjects and patients will be characterized. With all the variables obtained, network analyzes and predictive analyzes are carried out in order to see the interaction between variables and determine predictive variables of Alzheimer's disease that could be subject to modification by the diet. In a second stage, the personalized supplement will be designed based on the characteristics of Alzheimer's patients and there is no patient participation. In a third stage, a randomized, parallel nutritional intervention trial will be carried out where the supplement designed "ad hoc" will be compared in the population of Alzheimer's patients against a nutritional supplement commonly used in Alzheimer's patients.

ELIGIBILITY:
Inclusion Criteria:

1. to be able to give written consent signed jointly by the patient's legal representative following the rules of the clinical research ethics committee
2. minimum educational level (reading and writing)
3. proficiency of the language of the tests applied; adequate visual and auditory acuity, in the opinion of the researcher, to enable him/her to carry out the tests in the study (compensatory glasses and hearing aids are allowed
4. compliance with the diagnostic criteria of prodromal Alzheimer's Disease according to the criteria of the Institute on Aging- Alzheimer's Association [NIA-AA]: Global Deterioration Scale GDS≥ 2-3
5. Availability of a person ('caregiver') who has frequent and sufficient contact with the subject, so that he/she can provide precise information on the subject's day-to-day life, and attend the visits that are required by the study

Exclusion Criteria:

1. Suffer or have suffered from neurological (epilepsy, sleep disorders, etc.), psychiatric or any other type of pathology (sensory, hepatic, infectious, etc.) which, in the investigator's opinion, may affect their current cognition and functionality
2. Metabolic/endocrine disorders: Type I diabetes, the rest will not be excluded
3. Chronic or sporadic use of antibiotics, antifungals, antivirals or anti-parasitic agents and chronic use of proton pump inhibitors (omeprazole, etc.). The chronic medication that these patients take due to hypertension, diabetes, etc., should be recorded in the database but should not be a criterion for exclusion
4. Suffer from some type of pathology related to the gastrointestinal system or have undergone gastrointestinal surgery (ulcerative colitis, Crohn's disease, bariatric surgery)
5. Pre-menopause or perimenopause

Control patients: recruited among the relatives and companions of the patients and/or in primary care centers in the region of Murcia. The inclusion criteria for the control group will be the same as for the Alzheimer's group except for the requirements regarding cognitive impairment. The intention is for the control group to be similar in age and sex distribution to the Alzheimer's group.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiota | Baseline, an average of 1.5 years from baseline and change after three months
  1. Differences in fecal microbiota between healthy controls and Alzheimer's disease participants
  2. Changes in fecal microbiota in Alzheimer's disease participants before and after a nutritional intervention.
  Microbiota shotgun analysis

SECONDARY OUTCOMES:
Dietary habits characterization | Baseline, an average of 1.5 years from baseline and change after three months
  Diet characterization of healthy controls and Alzheimer's disease participants
  - Changes in diet in Alzheimer's disease participants before and after a nutritional intervention
  3-day registration questionnaire, a food consumption frequency questionnaire and adherence to mediterranean diet questionnaire will be used. Percentage of macronutrients ingested will be obtained.
Physical activity (PA) characterization | Baseline
  The International Physical Activity Questionnaire for Older People (IPAQ-E) quantifies subjects' activity in minutes per week and categorizes the results into Metabolic Equivalent of Task (MET) values. 1 MET is equivalent to 3.5 mL of oxygen consumed per kg per minute.
  PA is characterized as:
  Low: No PA is performed, or the activity is insufficient to reach moderate or high activity.
  Moderate: Involves three or more days of vigorous PA for at least 25 minutes per day, or five or more days of vigorous PA and/or walking for at least 30 minutes per day. Additionally, achieving an energy expenditure of at least 600 METs per minute per week through a combination of activities.
  High: Involves vigorous activity at least three days per week, resulting in an energy expenditure of 1500 METs per minute per week. Alternatively, seven or more days of a combination of walking, moderate, and/or vigorous activity, reaching an energy expenditure of at least 3000 METs per minute per week.
Blood lipopolysaccharide (LPS) | Baseline, an average of 1.5 years from baseline and change after three months
  Changes in LPS in healthy controls and Alzheimer's disease participants
  - Changes in LPS in Alzheimer's disease participants before and after a nutritional intervention
  To analyze circulating LPS levels in blood samples
Fecal Short chain fatty acids (SCFA) | Baseline, an average of 1.5 years from baseline and change after three months
  Changes in fecal SCFA in healthy controls and Alzheimer's disease participants
  - Changes in fecal SCFA in Alzheimer's disease participants before and after a nutritional intervention
  SCFA will be analyzed by High performance liquid chromatography (HPLC)
Metabolomic analysis | An average of 1.5 years from baseline and change after three months
  Changes in serum and fecal samples in Alzheimer's disease participants before and after a nutritional intervention to search for potential markers of the supplement's effect on health.
Bile fecal acids | Baseline, an average of 1.5 years from baseline and change after three months
  - Changes in fecal bile acids in Alzheimer's disease participants before and after a nutritional intervention Bile fecal acids will be analyzed by High performance liquid chromatography (HPLC)

CONTACTS AND LOCATIONS:
Overall Officials: Mar Larrosa, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (2):
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemente-Velasco S, de Lucas B, Tabone M, Bressa C, Gonzalez-Soltero MDR, Martinez-Lopez S, Bailen M, Dominguez-Balmaseda D, Castellanos N, Diez GG, Noguera-Perea F, Marin-Munoz J, Sanchez-Alonso P, Rey AI, Galvez BG, Larrosa M. Study protocol for design of a personalized dietary supplement based on the gut microbiota of Alzheimer's patients and evaluation of its effects in a pilot randomized controlled trial. Front Nutr. 2025 Sep 23;12:1653841. doi: 10.3389/fnut.2025.1653841. eCollection 2025. PMID 41064285